CLINICAL TRIAL: NCT03328442
Title: Evaluation of Patient Satisfaction After Root Coverage Procedure Using VISTA Technique Compared to Modified Coronally Advanced Flap Technique in Conjunction With Platelet Rich Fibrin-membrane.
Brief Title: Patient Satisfaction After Root Coverage Using VISTA Technique Compared to MCAF Technique With PRF.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Salah salaheldin, Assistant lecturer faculty of dentistry Nahda university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-10-30
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vista technique (Experimental): The vista technique with PRF membrane uses a Vestibular incision subperiosteal tunnel access in combination with Platelet rich fibrin membrane to treat gingival recession defects.
  Interventions: Procedure: VISTA Technique
- modified coronally advanced flap (Active Comparator): A modified coronally advanced flap utilising Platelet rich fibrin membrane to treat gingival recession defects.
  Interventions: Procedure: modified coronally advanced flap

INTERVENTIONS:
Procedure: VISTA Technique — VISTA with PRF membrane includes Treatment of recession class I and II using autologous PRF membrane
  Other Names: Vestibular incision subperiosteal tunnel access
  Arms: Vista technique
Procedure: modified coronally advanced flap — modified coronally advanced flap with PRF membrane for Treatment of recession class I and II
  Other Names: MCAF
  Arms: modified coronally advanced flap

SUMMARY:
VISTA technique with PRF compared to MCAF technique with PRF to treat gingival recession

DETAILED DESCRIPTION:
Comparison between two techniques for root coverage divided in two groups the first (test group) VISTA technique in conjunction with PRF-membrane and the second (control group)MCAF technique in conjunction with PRF-membrane for treating Miller's class I and II gingival recession defects.

Clinical Periodontal Records will be taken at baseline, 3 months and 6 months respectively.

Visual analogue scale for pain during one week after operation. Patient satisfaction record using questionnaire after 6 months.

ELIGIBILITY:
Inclusion Criteria:

- Age (18-55) Miller's classI and II multiple GR width of KG>2 mm

Exclusion Criteria:

* Systemic diseases Poor oral hygiene Smoking Patient allergy Miller's class III and IV

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | after 6 months
  Using a questionnaire which are designed in a dichotomous fashion (yes or no ) and calculated by percentage of answering yes.
  it not a scale, the following questions will be asked to the patients;
  1. did you feel pain in spite of the medication prescribed?
  2. did you perceive the course of healing unexpected restriction?
  3. did you experience any remaining symptoms of parasethesia?
  4. would you described the under taken effort as reasonable?
  5. have your expectations been fulfilled?

CONTACTS AND LOCATIONS:
Overall Officials: Azza Ezzelarab, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zadeh HH. Minimally invasive treatment of maxillary anterior gingival recession defects by vestibular incision subperiosteal tunnel access and platelet-derived growth factor BB. Int J Periodontics Restorative Dent. 2011 Nov-Dec;31(6):653-60. PMID 22140667
- [Background] Zucchelli G, De Sanctis M. Treatment of multiple recession-type defects in patients with esthetic demands. J Periodontol. 2000 Sep;71(9):1506-14. doi: 10.1902/jop.2000.71.9.1506. PMID 11022782
- [Background] Zuhr O, Rebele SF, Schneider D, Jung RE, Hurzeler MB. Tunnel technique with connective tissue graft versus coronally advanced flap with enamel matrix derivative for root coverage: a RCT using 3D digital measuring methods. Part I. Clinical and patient-centred outcomes. J Clin Periodontol. 2014 Jun;41(6):582-92. doi: 10.1111/jcpe.12178. Epub 2013 Nov 10. PMID 24117676